CLINICAL TRIAL: NCT04126356
Title: Evaluation of the Impact of the Sellick Manoeuvre or Para-tracheal Compression of the Cervical Esophagus on the Displacement of the Laryngeal Mass and the Visualization of the Vocal Cords
Brief Title: VIDEOLARYNGOSCOPY STUDY OF THE LPEC
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Other Study IDs: ANESBJ2019; 2019-001109-26 (EudraCT Number)
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Laryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mobilization of the larynx — Check the intubation conditions during laryngoscopy without external mobilization of the larynx, with Sellick manoeuvre or with low paratracheal esophagal compression.

SUMMARY:
Check the intubation conditions during laryngoscopy without external mobilization of the larynx, with Sellick manoeuvre or with low paratracheal esophagal compression.

DETAILED DESCRIPTION:
Check the intubation conditions during laryngoscopy without external mobilization of the larynx, with Sellick manoeuvre or with low paratracheal esophagal compression.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoing general anaesthesia

Exclusion Criteria:

* pregnant women
* people with facial
* oropharyngeal abnormalities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients undergoing general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Distance between oesophagus and trachea | During laryngoscopy procedure
  Distance between oesophagus and trachea

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, University Hospital, Liège, Belgium